CLINICAL TRIAL: NCT04479488
Title: Brazilian COVID-19 Registry for Clinical Presentation of Individuals With COVID-19: a National, Multicentre, Prospective Observational Study (SARS-Brazil)
Brief Title: Brazilian Registry for Clinical Presentation of Individuals With COVID-19 (SARS-Brazil)
Acronym: SARS-Brazil
Status: Completed | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: 30047620.3.0000.0071
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2022-12

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: COVID-19; SARS-CoV2 infection; Intensive care unit; Oxygen supplementation; Invasive ventilation; Mortality
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Blood, serum, plasma and nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalized patients: Patient who are suspected or confirmed SARS-CoV2 infection need hospitalization.
  Interventions: Other: Hospital admission
- Non-hospitalized patients: Patient who are suspected or confirmed SARS-CoV2 infection non-hospitalized.
  Interventions: Other: Non-hospitalization procedures

INTERVENTIONS:
Other: Hospital admission — Usual care.
  Groups: Hospitalized patients
Other: Non-hospitalization procedures — Usual care.
  Groups: Non-hospitalized patients

SUMMARY:
This is a registry-based cohort study of all adult patients (≥18 years) with confirmed or suspected SARS-CoV-2 infection.

The main goal is to describe mortality incidence, demographic characteristics, coexisting conditions, treatments, outcomes among SARS-CoV2 infected patients.

A secondary goal is to identify biological factors (OMICS - genomic, proteomic and metabolomics characterization) associated with severity conditions for these patients.

DETAILED DESCRIPTION:
Registry on characteristics and outcomes of hospitalized and non-hospitalized SARS-CoV2 infected patients in Brazil.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years);
* Confirmed or suspected SARS-CoV2 infection

Exclusion Criteria:

* Patient who expressed opposition to participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SARS-Brazil Registry is designed as multicenter observational cohort of adult patients (≥18 years old), that are confirmed or suspected SARS-CoV-2 infection in Brazilian hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1587 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 60 Days
  All-cause mortality rates at 60 days

SECONDARY OUTCOMES:
Incidence and course of symptoms of COVID-19 infection | 60 Days
  To assess the prevalence and course of symptoms of COVID-19 infection of patients followed during a period of 60 days
Hospitalizations | 60 Days
  Rate of patients requiring hospitalization and re-hospitalization (readmission to the hospital occurring within 60 days after admission)
Oxygen supplementation | 60 Days
  Rate of patients requiring oxygen therapy
Use of invasive mechanical ventilation | 60 Days
  Rate of patients requiring invasive mechanical ventilation
Intensive care unit length of stay | 60 Days
  ICU length of stay

OTHER OUTCOMES:
Serum proteomic | 60 Days
  Percentual changes in serum proteome of patients with mild or moderate to severe disease
Serum metabolomic | 60 Days
  Percentual changes in serum metabolome of patients with mild or moderate to severe disease
Genomic description | 60 Days
  Determination of whole genome sequence and transcriptomic of mild or moderate to severe disease

CONTACTS AND LOCATIONS:
Overall Officials: Otávio Berwanger, PhD, Study Director — Hospital Israelita Albert Einstein; Henrique A Fonseca, PhD, Principal Investigator — Hospital Israelita Albert Einstein
Locations (14):
- Brazil (14):
  - Hospital de Emergencia Dr. Daniel Houly, Arapiraca, Alagoas
  - Alencar Serviços Médicos Ltda, Barbalha, Ceará
  - Hospital Estadual Jayme dos Santos Neves, Serra, Espírito Santo
  - Hospital Santa Rita de Cássia, Vitória, Espírito Santo
  - Universidade Federal da Bahia, Vitória da Conquista, Estado de Bahia
  - Fundação Educacional Lucas Machado, Belo Horizonte, Minas Gerais
  - Fundação Hopitalar São Francisco de Assis, Belo Horizonte, Minas Gerais
  - Hospital Santa Lucia, Poços de Caldas, Minas Gerais
  - Hospital Giselda Trigueiro, Natal, Rio Grande do Norte
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
  - Hospital Municipal Vila Santa Catarina, São Paulo
  - Hospital São Camilo - Ipiranga, São Paulo
  - Hospital São Camilo - Pompéia, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fonseca HAR, Pereira AJ, Nawa RK, Sant'Anna VAR, Almeida TF, Guimaraes HP, Tognon AP, Marques LM, Silva LSCD, Bittencourt RS, Gomes CP, Martins PA, Oliveira AL, Milan EP, Dall'Orto FTC, Hoffman Filho CR, Almeida G, Hohmann FB, Moia DDF, Piano LPA, Machado FP, Soares RVP, Damiani LP, Assis SRL, Amaro Junior E, Rizzo LV, Berwanger O. Mortality, hospitalizations, and persistence of symptoms in the outpatient setting of the first COVID-19 wave in Brazil: results of SARS-Brazil cohort study. Einstein (Sao Paulo). 2024 Aug 9;22:eAO0652. doi: 10.31744/einstein_journal/2024AO0652. eCollection 2024. PMID 39140573